CLINICAL TRIAL: NCT03557034
Title: A Fib Clinic of the Future Using KardiaPro Platform for Chronic Care of Patients With AF After Ablation Procedure
Acronym: AliveCor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: AliveCor (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-444
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation
Keywords: pulmonary vein isolation; atrial fibrillation; remote monitoring; heart rhythm monitor
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care Monitoring (No Intervention): Standard of Care
- Kardia Monitoring (Experimental): Kardia Mobile/Kardia Pro
  Interventions: Device: Kardia Monitoring

INTERVENTIONS:
Device: Kardia Monitoring — Kardia Mobile is an FDA approved device that allows one lead ECG recording for 30 seconds using the patient's smart phone. The device has a built-in algorithm that detects AF. KardiaPro is a secure platform that allows the physician to access the patient's recording at any time. The platform can also be programmed to send a notification to the healthcare provider if AF is detected by the software.
  Arms: Kardia Monitoring

SUMMARY:
Pulmonary vein isolation is a widely used strategy for the treatment of patients with symptomatic atrial fibrillation. After successful pulmonary vein isolation (no atrial fibrillation on transtelephonic rhythm recordings for 3 months following ablation), heart rhythm is not routinely monitored. The goal of this study is to determine whether the Kardia Mobile device detects AF at a different rate compared to our standard of care. The study also hopes to understand how this Kardia Mobile device and Kardia Pro platform affect health care utilization and patient anxiety.

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) is a widely used strategy for the treatment of patients with symptomatic atrial fibrillation (AF). After ablation, patients are usually discharged with transtelephonic monitor. Patients are encouraged to send their electrophysiologist transmissions of their heart rhythm at least once a week or anytime they have symptoms. After 3-4 months of remote monitoring, patients come for their first visit after the ablation. At this visit, the electrophysiologist reviews the heart rhythm transmissions since the ablation and based on the findings, decisions are made regarding anticoagulation or antiarrhythmic drug therapy. If all transmissions show sinus rhythm and the patient is doing well, he or she is normally followed clinically based on symptoms without any rhythm monitors. Usually, these patients follow up in another 6 months with an ECG at the time of the visit with the caring electrophysiologist. During these 6 months, patients might experience palpitations or recurrent arrhythmias. These episodes usually trigger phone encounters with the provider and this can trigger additional testing. Sometimes it might lead to clinic or emergency room encounters.

Kardia Mobile is an FDA approved device that allows one lead ECG recording for 30 seconds using the patient's smart phone. The device has a built-in algorithm that detects AF. KardiaPro is a secure platform that allows the physician to access the patient's recording at any time. The platform can also be programmed to send a notification to the healthcare provider if AF is detected by the software. The goal of our study is to determine whether detection of AF with Kardia Mobile is different than the current standard approach and to assess the value of using Kardia Mobile and the KardiaPro platform in decreasing health care utilization and reducing patient anxiety following AF ablation.

ELIGIBILITY:
Inclusion Criteria:

1. 18-85 years old
2. Have smartphone with data plan
3. History of AF (paroxysmal or persistent)
4. In sinus rhythm at the 3-4 month post-procedure visit and no evidence of AF during the interval starting after the 3 week blanking period and ending at the appointment time.
5. On Anticoagulation if CHADS VASC score is ≥ 1 and will continue to be on anticoagulation or CHADS VASC of Zero
6. Willing to follow up with their Cleveland Clinic electrophysiologist in 6 months

Exclusion Criteria:

1. Patients without smartphone
2. Unwilling to provide consent
3. Unwilling to follow up in 6 months
4. CHADS VASC ≥ 1 and anticoagulation will be stopped
5. Presence of a cardiac implantable electronic device
6. If the primary electrophysiologist decides the patient still needs monitoring through traditional monitors due to any reason

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun G Tarajki, MD MPH, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Monitoring: Standard of Care: Patients will be followed clinically based on symptoms.
Period: Overall Study
Arm/Group | Standard of Care Monitoring | Kardia Monitoring
Started | 49 | 51
Randomization | 49 | 51
Completed | 48 | 51
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized patients that did not withdraw consent early
Groups:
- Standard of Care Monitoring: Standard of Care
  This is our current standard of care for following patients after successful AF ablation. Patients will be followed clinically based on symptoms (no monitor is provided). They will be seen for follow up 6 months after enrollment into the study. During these 6 months, patients can call if they have symptoms. The caring team will order any additional testing or monitors as deemed necessary by the patient's primary electrophysiologist. At the 6 months follow up visit with the patient's primary electrophysiologist, a 12 lead ECG is performed. The GAD7 will be administered at this visit.
- Total: Total of all reporting groups
Arm/Group | Standard of Care Monitoring | Kardia Monitoring | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (11.8) | 63.8 (8.5) | 64.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 35 | 35 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 44 | 51 | 95
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 51 | 99
Type of Afib at baseline [Count of Participants; unit: Participants]
  Paroxysmal | 23 | 26 | 49
  Persistent | 17 | 16 | 33
  Unknown | 8 | 9 | 17
CHADS-VASC score [Median (Inter-Quartile Range); unit: units on a scale] — CHA2DS2-VASc (congestive heart failure, hypertension, age ≥ 75 years, diabetes mellitus, stroke or transient ischemic attack, vascular disease, age 65 to 74 years, sex category) score is a validated tool to predict the risk of stroke and systemic emboli in patients with non-valvular atrial fibrillation. Score ranges 0 - 6. Oral anticoagulation is recommended for those patients with a score of 2 or greater, and oral anticoagulant or aspirin may be considered for a CHA2DS2-VASc score of 1.
  units on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Time to Atrial Fibrillation Detection
Description: This outcome will measure the time between the ablation procedure (time zero) and the time of first detected atrial fibrillation heart rhythm.
Time Frame: 6 months
Population: Randomized Patients that did not withdraw consent immediately
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care Monitoring | Kardia Monitoring
Number analyzed (Participants) | 48 | 51
days | 85.0 (62.8) | 77.6 (61.0)

2. Secondary Outcome: Incidence of Atrial Fibrillation After Successful AF Ablation
Description: Number (%) participants with Afib detected after ablation and during the study period.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Monitoring | Kardia Monitoring
Number analyzed (Participants) | 48 | 51
Participants | 7 | 11

3. Secondary Outcome: Number of Atrial Fibrillation Episodes Detected
Description: Number of abnormal reading using Kardia Mobile after ablation
Time Frame: 6 months
Population: Applies only to Kardia Mobile arm
Measure: Median (Inter-Quartile Range); unit: Number of abnormal reading
Arm/Group | Standard of Care Monitoring | Kardia Monitoring
Number analyzed (Participants) | 0 | 51
Number of abnormal reading |  | 11 [2 to 16]

4. Secondary Outcome: Average Number of Clinical Encounters After Successful Ablation
Description: Average number of phone encounters within 6 months after successful ablation
Time Frame: 6 months
Population: All randomized patients that did not withdraw consent immediately
Measure: Mean (Standard Deviation); unit: Number of phone encounters
Arm/Group | Standard of Care Monitoring | Kardia Monitoring
Number analyzed (Participants) | 48 | 51
Number of phone encounters | 2.9 (6.2) | 1.96 (2.7)

5. Secondary Outcome: Number of Participants Using Alternative Monitoring Devices After Successful Ablation
Description: Additional ECGs and ambulatory heart rhythm monitoring used (Holter, Ziopatch) during the follow up interval
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Monitoring | Kardia Monitoring
Number analyzed (Participants) | 48 | 51
Participants | 13 | 3

6. Secondary Outcome: Change in Level of Anxiety From the Date of Atrial Fibrillation Ablation to the End of Study Period
Description: The Generalized Anxiety Disorder-7 is a scale to measure the severity of anxiety. It consists of asking patients to respond to a simple questionnaire and each answer is assigned a point based on the frequency of a given symptom (0=Not at all, 1=Several days, 2= More than half the days, 3=Nearly everyday). Total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity. A total score of 5-9 indicates mild anxiety, 10-14 moderate anxiety, and >15 severe anxiety.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard of Care Monitoring | Kardia Monitoring
Number analyzed (Participants) | 48 | 51
units on a scale | -1.23 [-2.6 to 0.17] | 0.0 [-1.4 to 1.4]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Standard of Care Monitoring | Kardia Monitoring
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 0/48 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT03557034/Prot_SAP_000.pdf